CLINICAL TRIAL: NCT04658173
Title: A Randomized, Controlled Trial to Compare the Efficacy and Safety Profile of a Remimazolam-alfentanil Combination With a Propofol-alfentanil Combination for ERCP
Brief Title: Efficacy and Safety Profile of Remimazolam-alfentanil Combination for ERCP Sedation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Nankai Hospital (Other)
Responsible Party: Principal Investigator, Jianbo Yu, Director, Tianjin Nankai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NKYY_YXKT_IRB_2020_063_01
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Anesthesia
Keywords: ERCP; Propofol; Remimazolam; Alfentanil
MeSH Terms: interventions — clindamycin, tretinoin drug combination

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remimazolam-alfentanil combination (Experimental): Group remimazolam-alfentanil combination received 10 µg/kg alfentanil and 0.3mg/kg remimazolam over 30 seconds, followed by an infusion of remimazolam at 0.2 to 1 mg/kg/hr and alfentanil at 0 to 1ug/kg/min. In case of the sudden patient movement, and difficulty in maneuvering the endoscope, remimazolam 0.1mg/kg was used in the form of bolus, as rescue drugs, and alfentanil 5ug/kg when additional analgesia is needed
  Interventions: Drug: remimazolam-alfentanil combination
- propofol-alfentanil combination (Active Comparator): Group propofol-alfentanil combination received 10 µg/kg alfentanil and 1.5 to 2mg/kg propofol over 30 seconds followed by an infusion of propofol at 2 to 6 mg/kg/hr and alfentanil at 0 to 1ug/kg/min. In case of the sudden patient movement, and difficulty in maneuvering the endoscope, propofol 0.5 mg/kg was used in the form of bolus, as rescue drugs, and alfentanil 5ug/kg when additional analgesia is needed
  Interventions: Drug: propofol-alfentanil combination

INTERVENTIONS:
Drug: remimazolam-alfentanil combination — Group remimazolam-alfentanil combination received 10 µg/kg alfentanil and 0.3mg/kg remimazolam over 30 seconds, followed by an infusion of remimazolam at 0.2 to 1 mg/kg/hr and alfentanil at 0 to 1ug/kg/min. In case of the sudden patient movement, and difficulty in maneuvering the endoscope, remimazolam 0.1mg/kg was used in the form of bolus, as rescue drugs, and alfentanil 5ug/kg when additional analgesia is needed
  Other Names: RA Combination
  Arms: remimazolam-alfentanil combination
Drug: propofol-alfentanil combination — Group propofol-alfentanil combination received 10 µg/kg alfentanil and 1 mg/kg propofol over 30 seconds followed by an infusion of propofol at 2 to 6 mg/kg/hr. In case of the sudden patient movement, and difficulty in maneuvering the endoscope, propofol 0.5 mg/kg was used in the form of bolus, as rescue drugs，and alfentanil 5ug/kg when additional analgesia is needed
  Other Names: PA combination
  Arms: propofol-alfentanil combination

SUMMARY:
Moderate to deep levels of sedation and analgesia are required for ERCP. Propofol-based sedation is simple, easy to use, and effective, but is not without cardiovascular and respiratory adverse effects. The combination of remimazolam and alfentanil has shown promising results for sedation in other similar scenarios. The aim of this study was to compare the efficacy and safety of a standard propofol-alfentanil regimen with a remimazolam-alfentanil combination.

DETAILED DESCRIPTION:
What is already known about this topic is that propofol-based sedation techniques are effective for ERCP procedures but are not without cardiovascular and respiratory adverse effects.

1. Title:A randomized, controlled trial to compare the efficacy and safety profile of a remimazolam-alfentanil combination with a propofol-alfentanil combination for ERCP.
2. Research center: Single center.
3. The Design of the study: Randomized, double-blind, controlled study.
4. The population of the study: Age is between 18 and 85 years; ASA I-III levels; Patients undergone elective ERCP surgery, non-intubation patients;
5. Sample size: Based on Akhondzadeh R et al. research, propofol based sedation resulted in 43% patients present oxygen desaturation, and assuming a 15% reduction in hypoxic events in remimazolam group. From this, we have estimated that oxygen desaturation rate will be 43% in the propofol group and 28 % in the remimazolam group. We have estimated that, with a sample size of 207 patients, the study will have 80% power to detect a significant difference using the log-rank test. We have estimated that the rate of dropout or withdrawal will be approximately 20%, and thus we plan to enroll 259 patients each group
6. Interventions: Group remimazolam-alfentanil combination received 10 µg/kg alfentanil and 0.3mg/kg remimazolam over 30 seconds, followed by an infusion of remimazolam at 0.2 to 1 mg/kg/hr and alfentanil at 0 to 1ug/kg/min. In case of the sudden patient movement, and difficulty in maneuvering the endoscope, remimazolam 0.1mg/kg was used in the form of bolus, as rescue drugs, and alfentanil 5ug/kg when additional analgesia is needed.

   Group propofol-alfentanil combination received 10 µg/kg alfentanil and 1.5 to 2 mg/kg propofol over 30 seconds followed by an infusion of propofol at 2 to 6mg/kg/hr and alfentanil at 0 to 1ug/kg/min. In case of the sudden patient movement, and difficulty in maneuvering the endoscope,propofol 0.5mg/kg was used in the form of bolus, as rescue drugs, and alfentanil 5ug/kg when additional analgesia is needed.
7. Outcome： Primary outcome： The occurrence of hypoxia, defined by any event of SpO2 (oxygen saturation measured by pulse oximetry) < 90% of any duration.

   Secondary outcome： Number of events of hypoxia, defined as desaturation < 90%. The mean number of events during the procedure will be compared between the two groups.

   Lowest recorded SpO2 during the procedure. Requirement of minor airway manoeuvres: jaw lift/jaw thrust, nasopharyngeal airway insertion.

   Requirement of major airway manoeuvres: bag mask ventilation, endotracheal intubation.

   Total alfentanyl dose. The mean values (the doses in micrograms) during the procedure will be compared between the two groups.

   Requirement of antispasmodic agent. Proportion of patients requiring this medication will be compared between the two groups.

   Endoscope re-insertion rate. Rescued sedation: drugs dose. Total duration of procedure. Duration under sedation/anaesthesia. Successful completion of the procedure: Yes/No. Proportion of patients fulfilling this criterion will be compared between the two groups.

   Sensation of abdominal bloating: Y/N. Proportion of patients experiencing this adverse event will be compared between the two groups.

   Patients' satisfaction score on leaving recovery: 5 points numerical rating scale: Very satisfied (5), somewhat satisfied (4), neither satisfied nor dissatisfied (3), somewhat dissatisfied (2), very dissatisfied (1). Proportion of patients at a particular threshold will be compared between the two groups.

   The endoscopist assessed the ease of performing at the end of the procedure as I-satisfactory, II-difficult or III-impossible.

   QOR-15. Recovery time :The time to recovery based on Modified Aldrete score was noted every 5 minutes, starting from the time of endoscope removal . A score of 9 was considered as recovery and the patient was discharged to the ward.The estimated duration of the study:2-3 years.

   If the procure is expected more than 1 hour, the arterial blood gas (ABG) will be detected before and after the ERCP, and the serum Aβ1-40 will be also determined by the commercial kits.
8. Adverse events:

   Incidence of hypertention, hypotension，tachycardia , bradycardia，nausea，vomiting, POD, Sensation of abdominal bloating, The dosage of urapidil, ephedrine, atropine and esmolol during the observation period
9. Safety consideration: ECG, HR, MAP, respiratory rate was monitored.
10. Statistical analysis Mean and standard deviation values will be estimated for continuous outcomes while frequency and percentage will be computed for binary outcomes. 95% confidence intervals around the point estimate will be calculated where appropriate for the primary and secondary outcomes. Descriptive statistics will be used to present the results. P < 0.05 will be considered significant. Analyses will be intention-to-treat from randomisation. All randomised cases will be included in the analyses, regardless of missing data. As the data capture is only limited to a few hours after the intervention and the investigators are directly involved in the conduct of the study, we anticipate very few missing data. A subgroup analyses will be attempted (if feasible)

ELIGIBILITY:
Inclusion Criteria:

* Age is between 18 and 85 years
* ASA I-III levels;
* Patients undergone elective ERCP surgery, non-intubation patients;

Exclusion Criteria:

* Chronic pain with long-term use of analgesics, psychotropic substances (including opioids, NSAIDs, sedatives, antidepressants), alcohol abusers, with known drug allergy;
* BMI<18 or BMI>30;
* Abnormal renal function ;
* Previous abnormal surgical anesthesia recovery history;
* Hypertension or systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 95 mmHg when the patient admission to the operating room
* Sedatives, analgesics and antipruritic drugs were used 24 hours before operation;
* Expected difficult intubation ;
* Opioids allergy history;
* Take monoamine oxidase inhibitor or antidepressant within 15 days;
* Pregnant or parturient women;
* Involved in other drug trials within three months;
* Patients who can not communicate well with the researcher

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
The number of hypoxia | 1 day
  defined by any event of SpO2 (oxygen saturation measured by pulse oximetry) < 90% of any duration.

SECONDARY OUTCOMES:
Number of events of hypoxia, defined as desaturation < 90%. | 1 day
  The mean number of events during the procedure will be compared between the two groups
Lowest recorded SpO2 during the procedure | 1 day
  the lowest SpO2 during the procedure
the number of requirement for minor airway manoeuvres | 1 day
  such as jaw lift/jaw thrust, nasopharyngeal airway insertion.
the number of requirement for major airway manoeuvres | 1 day
  such as bag mask ventilation, endotracheal intubation.
Total alfentanyl dose | 1 day
  The mean values during the procedure will be compared between the two groups
Requirement of antispasmodic agent | 1 day
  Proportion of patients requiring this medication will be compared between the two groups
Endoscope re-insertion rate | 1 day
  Endoscope reinsertion
Rescued sedation: | 1 day
  drugs dose
Total duration of procedure | 1 day
  the duration of ERCP
Duration under sedation/anaesthesia | 1day
  Total anesthesia duration
Successful completion of the procedure | 1 day
  Yes/No. Proportion of patients fulfilling this criterion will be compared between the two groups
Sensation of abdominal bloating | 1-3 days
  Y/N. Proportion of patients experiencing this adverse event will be compared between the two groups
Patients' satisfaction score on leaving recovery | 1-3 days
  5 points numerical rating scale: Very satisfied (5), somewhat satisfied (4), neither satisfied nor dissatisfied (3), somewhat dissatisfied (2), very dissatisfied (1). Proportion of patients at a particular threshold will be compared between the two groups
The endoscopist assessed the ease of performing at the end of the procedure as I-satisfactory, II-difficult or III-impossible | 1 days
  The endoscopist assessed the ease of performing at the end of the procedure as I-satisfactory, II-difficult or III-impossible
quality of recovery score-15 | 1-3 days
  The quality of recovery score (QOR)-15 questionnaire
Recovery time | 1 day
  The time to recovery based on Modified Aldrete score was noted every 5 minutes, starting from the time of endoscope removal 9. A score of 9 was considered as recovery and the patient was discharged to the ward.

CONTACTS AND LOCATIONS:
Overall Officials: Jianbo Yu, MD, Principal Investigator — Tianjin Nankai Hospital
Locations (2):
- China (2):
  - Tianjin Nankai Hospital, Tianjin, Tianjin Municipality
  - Tianjin NanKai hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Akhondzadeh R, Ghomeishi A, Nesioonpour S, Nourizade S. A comparison between the effects of propofol-fentanyl with propofol-ketamine for sedation in patients undergoing endoscopic retrograde cholangiopancreatography outside the operating room. Biomed J. 2016 Apr;39(2):145-9. doi: 10.1016/j.bj.2015.11.002. Epub 2016 Jun 21. PMID 27372170
- [Result] Mazanikov M, Udd M, Kylanpaa L, Mustonen H, Lindstrom O, Farkkila M, Halttunen J, Poyhia R. A randomized comparison of target-controlled propofol infusion and patient-controlled sedation during ERCP. Endoscopy. 2013 Nov;45(11):915-9. doi: 10.1055/s-0033-1344712. Epub 2013 Oct 8. PMID 24104763
- [Result] Eberl S, Koers L, van Hooft J, de Jong E, Hermanides J, Hollmann MW, Preckel B. The effectiveness of a low-dose esketamine versus an alfentanil adjunct to propofol sedation during endoscopic retrograde cholangiopancreatography: A randomised controlled multicentre trial. Eur J Anaesthesiol. 2020 May;37(5):394-401. doi: 10.1097/EJA.0000000000001134. PMID 31860599
- [Result] Rex DK, Bhandari R, Desta T, DeMicco MP, Schaeffer C, Etzkorn K, Barish CF, Pruitt R, Cash BD, Quirk D, Tiongco F, Sullivan S, Bernstein D. A phase III study evaluating the efficacy and safety of remimazolam (CNS 7056) compared with placebo and midazolam in patients undergoing colonoscopy. Gastrointest Endosc. 2018 Sep;88(3):427-437.e6. doi: 10.1016/j.gie.2018.04.2351. Epub 2018 Apr 30. PMID 29723512
- [Result] Pastis NJ, Yarmus LB, Schippers F, Ostroff R, Chen A, Akulian J, Wahidi M, Shojaee S, Tanner NT, Callahan SP, Feldman G, Lorch DG Jr, Ndukwu I, Pritchett MA, Silvestri GA; PAION Investigators. Safety and Efficacy of Remimazolam Compared With Placebo and Midazolam for Moderate Sedation During Bronchoscopy. Chest. 2019 Jan;155(1):137-146. doi: 10.1016/j.chest.2018.09.015. Epub 2018 Oct 4. PMID 30292760
- [Result] Antonik LJ, Goldwater DR, Kilpatrick GJ, Tilbrook GS, Borkett KM. A placebo- and midazolam-controlled phase I single ascending-dose study evaluating the safety, pharmacokinetics, and pharmacodynamics of remimazolam (CNS 7056): Part I. Safety, efficacy, and basic pharmacokinetics. Anesth Analg. 2012 Aug;115(2):274-83. doi: 10.1213/ANE.0b013e31823f0c28. Epub 2011 Dec 20. PMID 22190555
- [Result] Goyal R, Hasnain S, Mittal S, Shreevastava S. A randomized, controlled trial to compare the efficacy and safety profile of a dexmedetomidine-ketamine combination with a propofol-fentanyl combination for ERCP. Gastrointest Endosc. 2016 May;83(5):928-33. doi: 10.1016/j.gie.2015.08.077. Epub 2015 Sep 11. PMID 26364968
- [Result] Thiruvenkatarajan V, Dharmalingam A, Arenas G, Wahba M, Steiner R, Kadam VR, Tran A, Currie J, Van Wijk R, Quail A, Ludbrook G. High-flow nasal cannula versus standard oxygen therapy assisting sedation during endoscopic retrograde cholangiopancreatography in high risk cases (OTHER): study protocol of a randomised multicentric trial. Trials. 2020 May 29;21(1):444. doi: 10.1186/s13063-020-04378-z. PMID 32471494
- [Result] Eberl S, Koers L, van Hooft JE, de Jong E, Schneider T, Hollmann MW, Preckel B. Sedation with propofol during ERCP: is the combination with esketamine more effective and safer than with alfentanil? Study protocol for a randomized controlled trial. Trials. 2017 Oct 11;18(1):472. doi: 10.1186/s13063-017-2197-8. PMID 29020995